CLINICAL TRIAL: NCT04318808
Title: Effect of Laser Acupuncture on Constipation in Patients With Advanced Cancer: a Prospective Double-blind Randomized Controlled Trial
Brief Title: Effect of Laser Acupuncture on Constipation in Patients With Advanced Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMRPG8K0031
Record Dates: First submitted 2020-03-16; First posted 2020-03-24 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2021-07

CONDITIONS: Constipation; Advanced Cancer
Keywords: Constipation; Acupuncture; Laser acupuncture; Advanced Cancer
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The participants in each group will receive real (with energy output) or sham (without energy output) laser acupuncture. The feelings of participants in each group are not different. The care provider and outcomes assessor don't involve the random allocation and don't know if participants receive real laser acupuncture.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LA group (Experimental): The subjects in the experimental group will receive 0.375 J of energy at each of the following acupoints: LI4 (Hegu, B3), LI11 (Quchi, B2), PC6 (Neiguan, B3), ST36 (Zusanli, B2), ST37 (Shangjuxu, B2), ST39 (Xiajuxu, B2), SP4 (Gongsun, B3) , SP9 (Yinlingquan, B2).
  Interventions: Procedure: Laser acupuncture
- Control group (Sham Comparator): The subjects in the control group will receive sham LA treatment, without any laser output (no stimulation) at the same acupoints used in experimental group.
  Interventions: Procedure: Laser acupuncture

INTERVENTIONS:
Procedure: Laser acupuncture — Laser acupuncture is a non-invasive therapy that involves stimulation of traditional acupoints with low-intensity, non-thermal laser irradiation.

SUMMARY:
Constipation is one of the most common complications in patients with advanced cancer.

The aim of this protocol designed as a double-blind randomized controlled trial is to investigate the efficacy of laser acupuncture (LA) therapy on constipation in patients with advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 years or older
* Principal diagnosis of advanced cancer
* Diagnosis of constipation
* Treat with laxatives for at least 1 week but still have symptoms of constipation

Exclusion Criteria:

* Intestinal obstruction
* Disturbance of consciousness
* Active gastrointestinal bleeding
* Active intraabdominal infection
* Local skin infection on the acupoints or limb amputees.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Complete spontaneous bowel movements (CSBM) | 1 week
  CSBM is defined as an spontaneous bowel movements associated with a sensation of complete evacuation. The number of CSBM within one week will be recorded.

SECONDARY OUTCOMES:
Comfort levels during defecation | 1 week
  Estimated using a 10-cm visual analogue scale with anchor points of 0 (no discomfort) and 10 (maximum discomfort).
Symptoms of constipation | 1 week
  A five-symptoms questionnaire for measuring the severity of constipation including straining during defecation, abdominal pain during defecation, hard stools, sensation of incomplete evacuation, and sensation of anorectal obstruction or blockage. Each item is rated on a four point Likert scale that ranges from severe symptom (4 points) to no symptom (1 point).
Colonic motility | 1 week
  Measured by auscultation of the lower right abdomen with a stethoscope.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Ting Liu, MD, Principal Investigator — Department of Chinese Medicine, Kaohsiung Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No